CLINICAL TRIAL: NCT06117215
Title: Prevalence of Premenstrual Syndrome in Women of Reproductive Age
Acronym: Sd-Premens
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Université de Reims Champagne-Ardenne (Other)
Responsible Party: Sponsor
Other Study IDs: 2023_RIPH_014_Sd-Premens
Record Dates: First submitted 2023-10-30; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Premenstrual Syndrome
Keywords: Premenstrual syndrome; women reproductive age; prevalence
MeSH Terms: conditions — Premenstrual Syndrome | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women of reproductive age: women of reproductive age
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — data collection

SUMMARY:
The menstrual cycle is a recurring process in the lives of women from puberty until menopause. This cycle can cause various discomforts, including premenstrual syndrome.

Described differently, premenstrual syndrome is a collection of physical and psychological symptoms that occur during the luteal phase of the menstrual cycle and subside upon the arrival of menstruation. This definition is conditioned by the existence of a free interval of at least one week between the end of the period and the appearance of these symptoms, as well as a global impairment of functioning and quality of life for women.

The impact on the personal, social, and professional lives of affected women, as well as the pain and discomfort it causes, may be perceived as insignificant or normal by women. Therefore, few women report the existence of these disorders to healthcare professionals. As the subject is not approached, these women are not taken care of even though therapeutic solutions could be proposed.

This pathology affects a large number of women, but its prevalence differs greatly depending on the studies conducted on the subject, suggesting a lack of knowledge of this syndrome.

DETAILED DESCRIPTION:
The main aim is to describe the prevalence of premenstrual syndrome among women of reproductive age.

ELIGIBILITY:
Inclusion Criteria:

* women in childbearing age, i.e., menstrual or secondary amenorrhoea, non-menopausal
* Over 18 years of age
* Agreeing to participate in the study

Exclusion Criteria:

* Menopause
* Having had a hysterectomy
* With primary amenorrhea
* Protected by law
* Refusing to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: women of chilbearing age
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
premenstrual syndrome | Day 0
  Prevalence of premenstrual syndrome defined as a set of physical, psychic and behavioral symptoms, appearing in the luteal phase of the menstrual cycle (that is, in the days before menstruation) and yielding with them, conditioned by a sufficient severity to alter the overall functioning and quality of life of women and must be present over at least 2 consecutive cycles.

CONTACTS AND LOCATIONS:
Overall Officials: Kristner Pauline, Dr, Principal Investigator — CH Épernay
Locations (1):
- Ufr Medecine Urca, Reims, France

IPD SHARING:
Plan to Share IPD: Undecided